CLINICAL TRIAL: NCT03900988
Title: A Randomized, Double Blind, Placebo Controlled Trial of Intravenous N-acetylcysteine and Oseltamivir Versus Intravenous 5% Dextrose and Oseltamivir in Adults Hospitalized With Influenza Complicated by Lower Respiratory Tract Infection.
Brief Title: Intravenous N-acetylcysteine and Oseltamivir Versus Oseltamivir in Adults Hospitalized With Influenza and Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAC Influenza/Hui/2019
Record Dates: First submitted 2019-03-31; First posted 2019-04-03 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Influenza
Keywords: respiratory, mortality, cytokines, chemokines, N-acetylcysteine (NAC)
MeSH Terms: conditions — Influenza, Human | interventions — Acetylcysteine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous N-acetylcysteine (NAC) and oseltamivir (Active Comparator)
  Interventions: Drug: N-acetyl cysteine
- intravenous 5% dextrose and oseltamivir (Placebo Comparator)
  Interventions: Drug: 5% Dextrose

INTERVENTIONS:
Drug: N-acetyl cysteine — N-acetyl cysteine will be administered at 100 mg/kg daily as a continuous IV infusion (in 1000ml of 5% dextrose) over 24 hrs and oseltamivir 75 mg bid orally for 5 days. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Arms: intravenous N-acetylcysteine (NAC) and oseltamivir
Drug: 5% Dextrose — 5% dextrose 1 liter given over 24 hrs and oral oseltamivir 75 mg bid for 5 days. Extension of dosing to 10 days for oseltamivir and the study drug is allowed if there is slow recovery, lack of improvement, or deterioration.
  Arms: intravenous 5% dextrose and oseltamivir

SUMMARY:
Seasonal influenza epidemics are important causes of morbidity and mortality. Cytokine dysregulation, with high levels of pro-inflammatory cytokines, occurs in patients with severe influenza. Early therapy with a neuraminidase inhibitor (NAI) is associated with better outcome in patients hospitalized with influenza, but significant mortality occurs despite use of antivirals. N-acetylcysteine (NAC) is a modified form of the amino acid cysteine, with anti-oxidant properties. NAC was shown to inhibit the production of pro-inflammatory molecules in lung epithelial cells infected with influenza viruses. Previous case report showed that high dose NAC, administered as continuous intravenous infusion, was effective and safe in improving the clinical outcomes. We aim to perform a randomized controlled trial to evaluate the therapeutic role of adjunctive NAC in the clinical management of patients with influenza complicated by lower respiratory tract involvement and abnormal respiratory status. Such information when available may reveal the potential of NAC for optimization of management of severe influenza, and provide important insights into future adjunctive therapy research.

ELIGIBILITY:
Inclusion Criteria:

* influenza A and B virus infections confirmed by polymerase chain reaction (PCR) and/or immunofluorescence assays,
* hospitalized for the management of severe manifestations of influenza,
* initiation of oseltamivir,
* clinical evidence of lower respiratory tract infection (e.g. shortness of breath, tachypnea, oxygen desaturation <93% on room air, crepitations on auscultation, infiltrations or consolidations on chest radiograph)
* written informed consent (by the subjects, or from their next of kin if the subjects are unable to provide written consent at the time of enrollment)

Exclusion Criteria:

* use of immunosuppressants (e.g. post-chemotherapy, post-transplant, autoimmune diseases) other than systemic corticosteroids
* known immuno-compromised conditions (e.g. active haematological malignancies, HIV/AIDS patients who are on antiretroviral therapy and CD4 cell count < 200),
* pregnancy
* lactation,
* end-stage renal failure
* hepatic failure
* cardiac failure
* patients on anticoagulation (except prophylactic dose of low molecular weight heparin),
* patients with scheduled major surgery within 2 weeks (NAC may affect blood clotting),
* patients who have received macrolide antibiotics and NSAID for 1 week prior to enrolment due to their immuno-modulating effects.
* Use of investigational anti-influenza antivirals and blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Normalization of respiratory status in day | 28 days
  oxygen saturation more than 93% or respiratory rate lower than 20/min on room air

SECONDARY OUTCOMES:
viral ribonucleic acid (RNA) in copies per milliliter | 28 days
  All serially collected samples will be subjected to viral ribonucleic acid (RNA) quantification using quantitative reverse transcription PCR (qRTPCR) targeting the matrix (M)-gene ('viral load')
Interleukin 6 in pg/ml | 10 days
interleukin-8 in pg/ml | 10 days
interleukin 17 in pg/ml | 10 days
Chemokine ligand 9 (CxCL9/MIG) in pg/ml | 10 days
Soluble tumour necrosis factor receptor-1 (sTNFR-1) in pg/ml | 10 days
interleukin 18 in pg/ml | 10 days
CRP in mg/L | 10 days
phospho-p38 and phospho-ERK (activated MAPKs) in mean fluorescence intensity(MFI) | 10 days
phospho-inhibitor kB/IkB (NF-kB) in mean fluorescence intensity(MFI) | 10 days
resolution of symptoms in days | 28 days
  A standard questionnaire will be used to collect baseline and serial clinical data. These include clinical manifestations/complications, symptom severity score, vital signs (e.g. temperature, respiratory rate, oxygen saturation), fever duration, requirements for supplemental oxygen therapy and invasive/non-invasive ventilation, duration of hospitalization, death, and occurrence of adverse events.
ICU admission in days | 28 days
mortality in days | 28 days
Incidence of Treatment-Emergent Adverse Events in numbers | 28 days
a six step ordinal scale of clinical status | 7 days
  death, in ICU, ongoing hospitalisation on oxygen, hospital stay not on oxygen, discharged but not returned to normal activities, or discharged and returned to normal activities

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No